CLINICAL TRIAL: NCT02548221
Title: The Assessment of Heart Function Using Transthoracic Echocardiogram (TTE) Following Thoracentesis on Large-volume Pleural Effusions
Brief Title: Impact of Large-Volume Pleural Effusions on Heart Function
Acronym: TTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Shi Huanzhong, Director of Department of Respiratory and Critical Care Medicine, Beijing Chaoyang Hospital, Beijing Chao Yang Hospital
Other Study IDs: TTE and LVPE
Record Dates: First submitted 2015-09-06; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Bilateral Pleural Effusion
Keywords: Thoracentesis; Pleural Effusions; Transthoracic echocardiogram; Lung volume measurements
MeSH Terms: conditions — Pleural Effusion | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: transthoracic echocardiogram — Thoracentesis was performed on patients with large-volume pleural effusions, and TTE was utilized to access the change of heart and lung function before and after this medical procedure.

SUMMARY:
The physiologic basis for relief from dyspnea after therapeutic thoracentesis remains poorly understood. Improvement of the heart and lung function may contribute to the dyspnea relief. But there is no data support this phenomenon. Transthoracic echocardiogram (TTE) is a non-invasive viewing of the heart, which can quickly assess the heart function through real-time images. The investigators performed thoracentesis on patients with large-volume pleural effusions, and utilized TTE to access the change of heart and lung function before and after this medical procedure.

DETAILED DESCRIPTION:
Patients with large pleural effusions often experience dramatic and immediate relief from dyspnea after therapeutic thoracentesis. Although this is a well-recognized phenomenon, the physiologic basis for such relief remains poorly understood. Primary physiologic basis for the relief in dyspnea after thoracentesis may include the improvement of the heart and lung function. In some cases the improvement in breathlessness cannot be attributed to the improvement of gas exchange, due to the atelectatic lung(not fully expansion of the lung). Transthoracic echocardiogram (TTE) is a non-invasive, real-time viewing of the internal parts of the heart using ultrasound, which can get highly accurate and quick assessment of the various heart images, though which doctors can quickly assess a patient's heart valves and degree of heart muscle contraction.

ELIGIBILITY:
Inclusion Criteria:

1. the estimated amount of effusion is above 500 ml;
2. Drainage was not performed within 1 month before admission;
3. assigned informed consent.

Exclusion Criteria:

1. physical weakness which is difficult to withstand the thoracentesis;
2. the happening of serious pleural reaction or reexpansion pulmonary edema on previous thoracentesis;
3. allergy to the anesthetic;
4. coagulation dysfunction, severe bleeding tendency;
5. serious mental illness who do not cooperate;
6. suspected with pleural hydatid disease;
7. skin infection around supine positioning;
8. severe heart function insufficiency who cannot lay on the back;
9. for a variety of reasons that cannot accept regular follow-up;
10. refused to sign the informed consent;
11. other conditions that is not suitable for the test.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with unilateral or bilateral pleural effusion, with at least 500ml amount of effusion are enrolled in this study. Study population include malignant pleural effusion, tuberculosis pleural effusion, parapneumonic effusion, and a variety of causes for transudative pleural effusion.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
changes of the TTE diameter after large-volume thoracentesis | baseline, immediately after drainage, 24 h after the thoracentesis
  change of the UCG diameter of the patients, including : Left ventricular: Left ventricular end-diastolic diameter(LVEDD）, Left ventricular end-systolic diameter（LVESD）, Left ventricular end-diastolic volume （LVEDV ）, Left ventricular end-systolic volume（ LVESV）, Left ventricular ejection fraction（LVEF）,Stroke volume（SV）,Cardiac output（CO），left ventricular diastolic function, including：E、A、E/A、E/Em、Em、Am（By PW&DTI）；Global longitudinal strain(GLS）; right ventricular：Basal and mid-cavity transversal right ventricular diameter, right ventricular free wall thickness, Tricuspid annular plane systolic excursion（TAPSE）, Fractional area change（FAC）, right ventricular systolic strain, Left and right atrial volume, coronary artery diameter

SECONDARY OUTCOMES:
changes of the distances on 6-MWT after large-volume thoracentesis | baseline, immediately after drainage, 24 h after the thoracentesis
  6-MWT is the distances on the 6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Huanzhong Shi, Ph.D, Study Director — Department of Respiratory and Critical Care Medicine, Beijing Chaoyang Hospital,
Locations (1):
- Department of Respiratory and Critical Care Medicine, Beijing Institute of Respiratory Medicine and Beijing Chaoyang Hospital, Capital Medical University, Beijing, China